CLINICAL TRIAL: NCT03500172
Title: An Adaptive Randomized Evaluation of Nurse-Led HIV Treatment Retention Interventions for Women Living With HIV in Durban, South Africa
Brief Title: HIV Treatment Retention Interventions for Women Living With HIV (Siyaphambili Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: University of the Western Cape (Other); TB HIV Care (Other); University of Toronto (Other); University of California, San Francisco (Other); National Institute for Communicable Diseases, South Africa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: R01NR016650 (NIH)
Record Dates: First submitted 2018-04-09; First posted 2018-04-17 (Actual); Results first posted 2023-09-21 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-12

CONDITIONS: HIV-1 Virologic Response
Keywords: HIV; Female Sex Workers; Viral Suppression; South Africa; Decentralized care; Antiretroviral therapy; Differentiated care

STUDY DESIGN:
Intervention Model Description: This sequential multistage adaptive randomized trial (SMART) assesses two interventions to address treatment barriers: (1) nurse-led mobile decentralized treatment programs (DTP) and (2) peer-led, individualized case management (ICM).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- DTP, Continue DTP if Responsive (Active Comparator): DTP:
  * Standard of care (SoC), minus clinic referrals for antiretroviral therapy (ART) treatment initiation and management.
  * Nurse initiated and managed ART within the community on mobile van at sites served by the mobile van which already provides SoC services
  Continues with DTP intervention if virally suppressed at 6 months.
  Interventions: Behavioral: DTP
- DTP, Standard of Care (SoC) if Responsive (Active Comparator): DTP:
  * Standard of care, minus clinic referrals for ART treatment initiation and management.
  * Nurse initiated and managed ART within the community on mobile van at sites served by the mobile van which already provides SoC services
  SoC:
  * HIV counseling and testing (HTC)
  * Sexually transmitted infection (STI) screening and treatment
  * Tuberculosis (TB) screening and referral
  * Health education through peer educators and peer supported follow-up related to linkages to care
  * Referrals to Department of Health (DoH) primary healthcare clinics or TB HIV Care (THC) drop-in center for ART treatment initiation and management
  Returns to SoC if virally suppressed at 6 months.
  Interventions: Behavioral: DTP
- DTP, Continue DTP if Non-Responsive (Active Comparator): DTP:
  * Standard of care, minus clinic referrals for ART treatment initiation and management.
  * Nurse initiated and managed ART within the community on mobile van at sites served by the mobile van which already provides SoC services
  Continues with DTP intervention if not virally suppressed at 6 months.
  Interventions: Behavioral: DTP
- DTP, DTP+ICM if Non-Responsive (Active Comparator): DTP:
  * Standard of care, minus clinic referrals for ART treatment initiation and management.
  * Nurse initiated and managed ART within the community on mobile van at sites served by the mobile van which already provides SoC services
  ICM:
  * Standard of Care
  * Assignment of peer case manager
  * Face-to-face meeting to tailor ICM approach to FSW preference
  * Self-efficacy building in face-to-face sessions and bi-weekly text messages
  * Relational support through monthly calls, face-to-face meetings every three months, and additional support through female sex worker (FSW) initiated interaction
  Receives both interventions at 6 months if non-virally suppressed.
  Interventions: Behavioral: DTP; Behavioral: ICM
- ICM, Continue ICM if Responsive (Active Comparator): ICM:
  * Standard of Care
  * Assignment of peer case manager
  * Face-to-face meeting to tailor ICM approach to FSW preference
  * Self-efficacy building in face-to-face sessions and bi-weekly text messages
  * Relational support through monthly calls, face-to-face meetings every three months, and additional support through FSW initiated interaction
  Continues with ICM intervention at 6 months if virally suppressed.
  Interventions: Behavioral: ICM
- ICM, SoC if Responsive (Active Comparator): ICM:
  * Standard of Care
  * Assignment of peer case manager
  * Face-to-face meeting to tailor ICM approach to FSW preference
  * Self-efficacy building in face-to-face sessions and bi-weekly text messages
  * Relational support through monthly calls, face-to-face meetings every three months, and additional support through FSW initiated interaction
  SoC:
  * HIV counseling and testing (HTC)
  * STI screening and treatment
  * TB screening and referral
  * Health education through peer educators and peer supported follow-up related to linkages to care
  * Referrals to DOH primary healthcare clinics or THC drop-in center for ART treatment initiation and management
  Returns to SoC if virally suppressed at 6 months.
  Interventions: Behavioral: ICM
- ICM, Continue ICM if Non-Responsive (Active Comparator): ICM:
  * Standard of Care
  * Assignment of peer case manager
  * Face-to-face meeting to tailor ICM approach to FSW preference
  * Self-efficacy building in face-to-face sessions and bi-weekly text messages
  * Relational support through monthly calls, face-to-face meetings every three months, and additional support through FSW initiated interaction
  Continues with ICM intervention at 6 months if non-virally suppressed.
  Interventions: Behavioral: ICM
- ICM, ICM+DTP if Non-Responsive (Active Comparator): ICM:
  * Standard of Care
  * Assignment of peer case manager
  * Face-to-face meeting to tailor ICM approach to FSW preference
  * Self-efficacy building in face-to-face sessions and bi-weekly text messages
  * Relational support through monthly calls, face-to-face meetings every three months, and additional support through FSW initiated interaction
  DTP:
  * Standard of care, minus clinic referrals for ART treatment initiation and management.
  * Nurse initiated and managed ART within the community on mobile van at sites served by the mobile van which already provides SoC services
  Receives both interventions at 6 months if non-virally suppressed.
  Interventions: Behavioral: DTP; Behavioral: ICM
- Standard of Care (SoC) (No Intervention): Standard of Care (SoC):
  * HIV counseling and testing (HTC)
  * Sexually transmitted infection (STI) screening and treatment
  * Tuberculosis (TB) screening and referral
  * Health education through peer educators and peer supported follow-up related to linkages to care
  * Referrals to Department of Health (DoH) primary healthcare clinics or TB HIV Care (THC) drop-in center for ART treatment initiation and management

INTERVENTIONS:
Behavioral: DTP — Provision of antiretroviral therapy (ART) in the community through a mobile-van DTP managed by a nurse capable of initiating and managing ART.
  Arms: DTP, Continue DTP if Non-Responsive; DTP, Continue DTP if Responsive; DTP, DTP+ICM if Non-Responsive; DTP, Standard of Care (SoC) if Responsive; ICM, ICM+DTP if Non-Responsive
Behavioral: ICM — Peer-led ICM through quarterly face-to-face meetings, monthly phone calls and biweekly text messages.
  Arms: DTP, DTP+ICM if Non-Responsive; ICM, Continue ICM if Non-Responsive; ICM, Continue ICM if Responsive; ICM, ICM+DTP if Non-Responsive; ICM, SoC if Responsive

SUMMARY:
The Siyaphambili Study is a sequential multistage adaptive randomized trial (SMART) to compare the effectiveness and durability of two behavioral interventions on the HIV-1 virologic response among female sex workers (FSW) living with HIV in Durban, South Africa. The interventions are: 1) nurse-led decentralized treatment program (DTP) and 2) individualized case management (ICM). Viral suppression is defined as a viral load assessment <50 RNA copies/mL. The design will also estimate the incremental cost-effectiveness of study interventions and combinations of interventions compared with maintaining the South African standard of HIV care and treatment.

DETAILED DESCRIPTION:
RATIONALE: Approximately 60% of the estimated 121,000 - 167,000 female sex workers (FSW) in South Africa are living with HIV. Research suggests only 39% of these women are currently on antiretroviral therapy (ART) and face individual, network and structural level barriers to ART initiation, retention and adherence. To prevent clinical treatment outcome disparities and reduce onward HIV transmission, understanding how best to adapt and implement, scalable and effective interventions to promote viral suppression among marginalized women is paramount. The overall goal of the Siyaphambili study is to inform South African HIV service delivery and scale up determining the most cost-effective package needed to achieve viral suppression among FSW and by characterizing the FSW most in need of these intensive HIV treatment interventions.

HYPOTHESIS: DTP and ICM will be equally effective at achieving viral suppression and will have a synergistic effect when combined and targeted at those who remain non-responsive to either isolated intervention. Additionally, an adaptive, graduated multicomponent intervention to achieve viral suppression would be preferred under standard thresholds for cost-effectiveness over single-intensity interventions or intensive multicomponent interventions for all FSW.

INTERVENTION: The Siyaphambili Study is a sequential multistage adaptive randomized trial (SMART) to compare the effectiveness and durability of two behavioral interventions on the HIV-1 virologic response among FSW living with HIV in Durban, South Africa. The interventions are: 1) nurse-led decentralized treatment program (DTP) and 2) individualized case management (ICM). The design will also estimate the incremental cost-effectiveness of study interventions and combinations of interventions compared with maintaining the South African standard of HIV care and treatment.

STUDY DESIGN: A sequential multistage adaptive randomized study, embedded within the TB/HIV Care program in Durban, South Africa, will enroll 800 viremic FSW into the 18-month trial. Women will be randomized to either DTP or ICM at enrolment and rerandomized 6 months after enrolment based on their response to the initial intervention.

PRIMARY OBJECTIVE: To compare the effectiveness and durability of nurse-led DTP and ICM in isolation or in combination to achieve viral suppression.

SECONDARY OBJECTIVE: To estimate the incremental impact and cost-effectiveness associated with study interventions and combination of interventions.

OUTCOMES: The primary outcome of the study is retention and viral suppression among those initially randomized to the DTP verse ICM intervention. The secondary outcomes are retention and viral suppression of non-responders, retention and viral suppression among month 6 non-responders, retention and viral suppression at 18 months among month 6 non-responders randomized to continuation of either intervention verse combined DTP+ICM, risk stratification tool, durability of retention and viral suppression of responders, to assess adherence, to assess viral suppression of retained, loss-to-follow-up, intervention acceptability, switching to 2nd/3rd line ART, and ART resistance.

ANALYTIC PLAN:

Primary analysis for primary outcome:

Retention in ART care and viral suppression will be a combined outcome in an intention to treat (ITT) analysis at 18 months to compare participants initially randomized to the DTP verse ICM intervention. Viral suppression is defined as a viral load assessment <50 RNA copies/mL and participants lost to follow up or who experience death during the trial duration will be grouped with non-virally suppressed participants.

ELIGIBILITY:
Inclusion Criteria:

1. Sells sex for goods or money as their main source of income
2. Assigned female sex at birth
3. ≥ 18 years of age
4. Living with HIV; diagnosed ≥ 6 months prior
5. Currently living in Durban
6. If on ART, initiated ≥2 months prior

Exclusion Criteria:

1. Engagement in an ongoing HIV treatment research study
2. Planning on leaving Durban for more than 3 months in the following 12 months
3. Pregnant at time of enrollment
4. On a second line or third ART regimen
5. Participating in an adherence club

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only cisgender women will be enrolled into the study.
Enrollment: 1391 (Actual)
Dates: Start 2018-06-22 (Actual); Primary Completion 2021-11-24 (Actual); Study Completion 2022-01-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Baral, MD, MPH, Principal Investigator — Johns Hopkins Bloomberg School of Public Health; Harry Hausler, MD, MPH, Principal Investigator — TB HIV Care
Locations (1):
- TB HIV Care, Durban, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Comins CA, Genberg B, Mcingana M, Bandeen-Roche K, Phetlhu DR, Steingo J, Mishra S, Wang L, Baral S, Hausler H, Schwartz S. Longitudinal Trajectories of Engagement With HIV Treatment Support Strategies Among Female Sex Workers Living With HIV in South Africa. J Acquir Immune Defic Syndr. 2025 Dec 1;100(4):323-330. doi: 10.1097/QAI.0000000000003738. PMID 40810449
- [Derived] Comins CA, Baral S, Mcingana M, Shipp L, Phetlhu DR, Young K, Guddera V, Hausler H, Schwartz S. ART coverage and viral suppression among female sex workers living with HIV in eThekwini, South Africa: Baseline findings from the Siyaphambili study. PLOS Glob Public Health. 2024 May 22;4(5):e0002783. doi: 10.1371/journal.pgph.0002783. eCollection 2024. PMID 38776334
- [Derived] Bhardwaj A, Comins CA, Guddera V, Mcingana M, Young K, Phetlhu R, Mulumba N, Mishra S, Hausler H, Baral S, Schwartz S. Prevalence of depression, syndemic factors and their impact on viral suppression among female sex workers living with HIV in eThekwini, South Africa. BMC Womens Health. 2023 May 5;23(1):232. doi: 10.1186/s12905-023-02392-2. PMID 37147708
- [Derived] Chen C, Baral S, Comins CA, Mcingana M, Wang L, Phetlhu DR, Mulumba N, Guddera V, Young K, Mishra S, Hausler H, Schwartz SR. HIV- and sex work-related stigmas and quality of life of female sex workers living with HIV in South Africa: a cross-sectional study. BMC Infect Dis. 2022 Dec 6;22(1):910. doi: 10.1186/s12879-022-07892-4. PMID 36474210
- [Derived] Wang L, Dowdy DW, Comins CA, Young K, Mcingana M, Mulumba N, Mhlophe H, Chen C, Hausler H, Schwartz SR, Baral S, Mishra S; Siyaphambili Study team. Health-related quality of life of female sex workers living with HIV in South Africa: a cross-sectional study. J Int AIDS Soc. 2022 Feb;25(2):e25884. doi: 10.1002/jia2.25884. PMID 35212470

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place at sex work venues and the TB HIV Care drop-in center in Durban, South Africa from June 2018 to March 2020. The first participant was enrolled on June 22, 2018 and the last participant was enrolled on March 23, 2020.
Pre-assignment Details: Of the 1391 participants enrolled, 777 met randomization criteria (non-virally suppressed) and were randomized to one of the two tested strategies. Participants who were virally suppressed at baseline OR lost to follow up prior to baseline randomization (n=614) continued with standard of care and were not randomized.
Groups:
- DTP, Continue DTP if Responsive: DTP:
  * Standard of care, minus clinic referrals for ART treatment initiation and management.
  * Nurse initiated and managed ART within the community on mobile van at sites served by the mobile van which already provides SoC services
  Continues with DTP intervention if virally suppressed at 6 months.
  DTP: Provision of antiretroviral therapy (ART) in the community through a mobile-van DTP managed by a nurse capable of initiating and managing ART.
- DTP, Standard of Care (SoC) if Responsive: DTP:
  * Standard of care, minus clinic referrals for ART treatment initiation and management.
  * Nurse initiated and managed ART within the community on mobile van at sites served by the mobile van which already provides SoC services
  SoC:
  * HIV counseling and testing (HTC)
  * STI screening and treatment
  * TB screening and referral
  * Health education through peer educators and peer supported follow-up related to linkages to care
  * Referrals to DOH primary healthcare clinics or THC drop-in center for ART treatment initiation and management
  Returns to SoC if virally suppressed at 6 months.
  DTP: Provision of antiretroviral therapy (ART) in the community through a mobile-van DTP managed by a nurse capable of initiating and managing ART.
- DTP, Continue DTP if Non-Responsive: DTP:
  * Standard of care, minus clinic referrals for ART treatment initiation and management.
  * Nurse initiated and managed ART within the community on mobile van at sites served by the mobile van which already provides SoC services
  Continues with DTP intervention if not virally suppressed at 6 months.
  DTP: Provision of antiretroviral therapy (ART) in the community through a mobile-van DTP managed by a nurse capable of initiating and managing ART.
- DTP, DTP+ICM if Non-Responsive: DTP:
  * Standard of care, minus clinic referrals for ART treatment initiation and management.
  * Nurse initiated and managed ART within the community on mobile van at sites served by the mobile van which already provides SoC services
  Receives both interventions at 6 months if non-virally suppressed.
  DTP: Provision of antiretroviral therapy (ART) in the community through a mobile-van DTP managed by a nurse capable of initiating and managing ART.
  ICM: Peer-led ICM through quarterly face-to-face meetings, monthly phone calls and biweekly text messages.
- ICM, Continue ICM if Responsive: ICM:
  * Standard of Care
  * Assignment of peer case manager
  * Face-to-face meeting to tailor ICM approach to FSW preference
  * Self-efficacy building in face-to-face sessions and bi-weekly text messages
  * Relational support through monthly calls, face-to-face meetings every three months, and additional support through FSW initiated interaction
  Continues with ICM intervention at 6 months if virally suppressed.
  ICM: Peer-led ICM through quarterly face-to-face meetings, monthly phone calls and biweekly text messages.
- ICM, SoC if Responsive: ICM:
  * Standard of Care
  * Assignment of peer case manager
  * Face-to-face meeting to tailor ICM approach to FSW preference
  * Self-efficacy building in face-to-face sessions and bi-weekly text messages
  * Relational support through monthly calls, face-to-face meetings every three months, and additional support through FSW initiated interaction
  SoC:
  * HIV counseling and testing (HTC)
  * STI screening and treatment
  * TB screening and referral
  * Health education through peer educators and peer supported follow-up related to linkages to care
  * Referrals to DOH primary healthcare clinics or THC drop-in center for ART treatment initiation and management
  Returns to SoC if virally suppressed at 6 months.
  ICM: Peer-led ICM through quarterly face-to-face meetings, monthly phone calls and biweekly text messages.
- ICM, Continue ICM if Non-Responsive: ICM:
  * Standard of Care
  * Assignment of peer case manager
  * Face-to-face meeting to tailor ICM approach to FSW preference
  * Self-efficacy building in face-to-face sessions and bi-weekly text messages
  * Relational support through monthly calls, face-to-face meetings every three months, and additional support through FSW initiated interaction
  Continues with ICM intervention at 6 months if non-virally suppressed.
  ICM: Peer-led ICM through quarterly face-to-face meetings, monthly phone calls and biweekly text messages.
- ICM, ICM+DTP if Non-Responsive: ICM:
  * Standard of Care
  * Assignment of peer case manager
  * Face-to-face meeting to tailor ICM approach to FSW preference
  * Self-efficacy building in face-to-face sessions and bi-weekly text messages
  * Relational support through monthly calls, face-to-face meetings every three months, and additional support through FSW initiated interaction
  DTP:
  * Standard of care, minus clinic referrals for ART treatment initiation and management.
  * Nurse initiated and managed ART within the community on mobile van at sites served by the mobile van which already provides SoC services
  Receives both interventions at 6 months if non-virally suppressed.
  DTP: Provision of antiretroviral therapy (ART) in the community through a mobile-van DTP managed by a nurse capable of initiating and managing ART.
  ICM: Peer-led ICM through quarterly face-to-face meetings, monthly phone calls and biweekly text messages.
- Standard of Care (SoC): SoC (virally suppressed at baseline OR lost to follow up prior to baseline randomization):
  * HIV counseling and testing (HTC)
  * STI screening and treatment
  * TB screening and referral
  * Health education through peer educators and peer supported follow-up related to linkages to care
  * Referrals to DOH primary healthcare clinics or THC drop-in center for ART treatment initiation and management
- Baseline Randomization: ICM: ICM:
  * Standard of Care
  * Assignment of peer case manager
  * Face-to-face meeting to tailor ICM approach to FSW preference
  * Self-efficacy building in face-to-face sessions and bi-weekly text messages
  * Relational support through monthly calls, face-to-face meetings every three months, and additional support through FSW initiated interaction
- Baseline Randomization: DTP: DTP:
  * Standard of care, minus clinic referrals for ART treatment initiation and management.
  * Nurse initiated and managed ART within the community on mobile van at sites served by the mobile van which already provides SoC services
Period: Period 1: Baseline Randomization
Arm/Group | DTP, Continue DTP if Responsive | DTP, Standard of Care (SoC) if Responsive | DTP, Continue DTP if Non-Responsive | DTP, DTP+ICM if Non-Responsive | ICM, Continue ICM if Responsive | ICM, SoC if Responsive | ICM, Continue ICM if Non-Responsive | ICM, ICM+DTP if Non-Responsive | Standard of Care (SoC) | Baseline Randomization: ICM | Baseline Randomization: DTP
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 614 | 390 | 387
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 614 | 387 | 387
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Period: Period 2: Re-Randomization
Arm/Group | DTP, Continue DTP if Responsive | DTP, Standard of Care (SoC) if Responsive | DTP, Continue DTP if Non-Responsive | DTP, DTP+ICM if Non-Responsive | ICM, Continue ICM if Responsive | ICM, SoC if Responsive | ICM, Continue ICM if Non-Responsive | ICM, ICM+DTP if Non-Responsive | Standard of Care (SoC) | Baseline Randomization: ICM | Baseline Randomization: DTP
Started | 27 | 24 | 171 | 165 | 20 | 27 | 177 | 163 | 614 | 0 | 0
Completed | 19 | 18 | 84 | 93 | 14 | 21 | 109 | 87 | 614 | 0 | 0
Not Completed | 8 | 6 | 87 | 72 | 6 | 6 | 68 | 76 | 0 | 0 | 0
Not completed — Lost to Follow-up | 8 | 6 | 87 | 68 | 4 | 6 | 63 | 74 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 4 | 2 | 0 | 5 | 2 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Non-virally suppressed participants who not lost to follow up prior to baseline randomization were randomized into two arms at baseline, DTP or ICM, presented here. Virally suppressed at baseline participants and non-virally suppressed participants who were lost to follow up prior to baseline randomization received standard of care.
Groups:
- Individualized Case Management (ICM) at Baseline: ICM:
  * Standard of Care
  * Assignment of peer case manager
  * Face-to-face meeting to tailor ICM approach to FSW preference
  * Self-efficacy building in face-to-face sessions and bi-weekly text messages
  * Relational support through monthly calls, face-to-face meetings every three months, and additional support through FSW initiated interaction
- Decentralized Treatment Provision (DTP) at Baseline: DTP:
  * Standard of care (SoC), minus clinic referrals for antiretroviral therapy (ART) treatment initiation and management.
  * Nurse initiated and managed ART within the community on mobile van at sites served by the mobile van which already provides SoC services
- Standard of Care (Virally Suppressed at Baseline OR Lost to Follow up Before Baseline Randomization): SoC (virally suppressed at baseline OR lost to follow up prior to baseline randomization):
  * HIV counseling and testing (HTC)
  * STI screening and treatment
  * TB screening and referral
  * Health education through peer educators and peer supported follow-up related to linkages to care
  * Referrals to DOH primary healthcare clinics or THC drop-in center for ART treatment initiation and management
- Total: Total of all reporting groups
Arm/Group | Individualized Case Management (ICM) at Baseline | Decentralized Treatment Provision (DTP) at Baseline | Standard of Care (Virally Suppressed at Baseline OR Lost to Follow up Before Baseline Randomization) | Total
Number analyzed (Participants) | 390 | 387 | 614 | 1391
Age, Customized [Count of Participants; unit: Participants]
  Age: 18-24 | 60 | 64 | 78 | 202
  Age: 25-29 | 135 | 123 | 119 | 377
  Age: 30-35 | 113 | 117 | 172 | 402
  Age: 35+ | 82 | 82 | 240 | 404
  Age: Missing | 0 | 1 | 5 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 390 | 387 | 614 | 1391
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 375 | 372 | 594 | 1341
  White | 0 | 0 | 0 | 0
  More than one race | 13 | 12 | 10 | 35
  Unknown or Not Reported | 2 | 1 | 9 | 12
Region of Enrollment [Count of Participants; unit: Participants]
  South Africa | 390 | 387 | 614 | 1391
Nationality [Count of Participants; unit: Participants]
  South African | 379 | 380 | 595 | 1354
  Other (Incl. Lesotho, Eswatini, Zimbabwe, Botswana) | 11 | 7 | 19 | 37
Education [Count of Participants; unit: Participants]
  Never attended | 4 | 6 | 15 | 25
  Complete/incomplete primary education | 29 | 28 | 79 | 136
  Secondary school incomplete | 283 | 278 | 394 | 955
  Secondary school complete | 54 | 67 | 98 | 219
  Any post-secondary education or technical training | 18 | 7 | 19 | 44
  Missing | 2 | 1 | 9 | 12
Currently enrolled in school [Count of Participants; unit: Participants]
  Currently enrolled in school | 2 | 1 | 9 | 12
  Not currently enrolled in school | 388 | 386 | 605 | 1379
Can read and/or write in Zulu or English [Count of Participants; unit: Participants] | 382 | 379 | 585 | 1346
Current employment other than sex work [Count of Participants; unit: Participants]
  None | 371 | 366 | 561 | 1298
  Self-employed (formal or informal) | 14 | 16 | 33 | 63
  Private or public employed | 2 | 3 | 10 | 15
  Refusal | 0 | 1 | 0 | 1
  Missing | 3 | 1 | 10 | 14
Relationship status [Count of Participants; unit: Participants]
  Steady partner, living together | 59 | 64 | 86 | 209
  Steady partner, not living together | 116 | 134 | 221 | 471
  Single | 213 | 188 | 298 | 699
  Missing | 2 | 1 | 9 | 12
Median age at first sex [Median (Inter-Quartile Range); unit: years] | 16 [15 to 18] | 17 [15 to 18] | 17 [15 to 18] | 17 [15 to 18]
Median age at first exchange of sex acts for goods [Median (Inter-Quartile Range); unit: years] | 22 [20 to 26] | 22 [19 to 25] | 23 [20 to 28] | 22 [20 to 27]
Median age at first exchange of sex acts for money [Median (Inter-Quartile Range); unit: years] | 22 [20 to 27] | 22 [20 to 26] | 23 [20 to 28] | 23 [20 to 27]
Advertises service online [Count of Participants; unit: Participants] | 15 | 10 | 29 | 54
Always carries condoms while working [Count of Participants; unit: Participants] | 341 | 333 | 529 | 1203
Consistent condom use with new clients (last 30 days) [Count of Participants; unit: Participants]
  Consistent | 223 | 226 | 371 | 820
  Inconsistent | 145 | 146 | 210 | 501
  Refusal/missing | 10 | 7 | 15 | 32
  Did not have sex with a new client in last 30 days | 12 | 8 | 18 | 38
Consistent condom use with regular clients (last 30 days) [Count of Participants; unit: Participants]
  Consistent | 183 | 186 | 312 | 681
  Inconsistent | 179 | 174 | 260 | 613
  Refusal/missing | 11 | 7 | 17 | 35
  Did not have sex with a regular client in the last 30 days | 17 | 20 | 25 | 62
Consistent condom use with non-paying partners (last 30 days) [Count of Participants; unit: Participants]
  Consistent | 55 | 37 | 77 | 169
  Inconsistent | 138 | 165 | 256 | 559
  No sex with non-paying partner in past 30 days | 190 | 182 | 264 | 636
  Refusal/missing | 7 | 3 | 17 | 27
Hormonal contraception [Count of Participants; unit: Participants] | 130 | 119 | 236 | 485
Non-hormonal contraception [Count of Participants; unit: Participants] | 378 | 377 | 588 | 1343
Parity [Count of Participants; unit: Participants]
  Nulliparous/No live births | 90 | 83 | 105 | 278
  One live birth | 136 | 136 | 182 | 454
  Two live births | 96 | 86 | 142 | 324
  Three or more live births | 68 | 81 | 183 | 332
  Missing | 0 | 1 | 2 | 3
Tested for tuberculosis in last 6 months [Count of Participants; unit: Participants] | 224 | 227 | 374 | 825
Hospitalized in last 6 months [Count of Participants; unit: Participants] | 40 | 40 | 76 | 156
Antiretroviral therapy experience [Count of Participants; unit: Participants]
  ART Naive | 70 | 72 | 37 | 179
  Ever Initiated | 320 | 315 | 573 | 1208
  Missing | 0 | 0 | 4 | 4
Ever experienced physical abuse [Count of Participants; unit: Participants] | 231 | 215 | 297 | 743
Ever experienced sexual abuse [Count of Participants; unit: Participants] | 159 | 166 | 192 | 517
Median self-reported health state [Median (Inter-Quartile Range); unit: units on a scale] — This measure uses a Median Self-reported Health Scale which ranges from 0 to 100. Participants were asked to respond to the following prompt: "To help people say how good or bad a health state is, we have drawn a scale (rather like a thermometer) on which the best state you can imagine is marked 100 and the worst state you can imagine is marked 0. We would like you to indicate on this scale how good or bad your health is today, in your opinion."
  units on a scale | 51 [44 to 66] | 51 [47 to 70] | 56 [50 to 75] | 52 [50 to 70]
Depression [Count of Participants; unit: Participants]
  No/minimal depression | 66 | 78 | 114 | 258
  Mild depression | 178 | 176 | 287 | 641
  Moderate depression | 47 | 52 | 89 | 188
  Moderately severe depression | 72 | 54 | 67 | 193
  Severe depression | 22 | 22 | 37 | 81
  Missing | 5 | 5 | 20 | 30
Drinks alcohol two or more times a week [Count of Participants; unit: Participants] | 165 | 163 | 240 | 568
Ever injected drugs [Count of Participants; unit: Participants] | 23 | 21 | 13 | 57
Baseline viral load [Count of Participants; unit: Participants]
  Less than 50 copies/mL (virally suppressed) | 0 | 0 | 523 | 523
  50 to 1000 copies/mL (non-virally suppressed) | 96 | 87 | 28 | 211
  Greater than 1000 copies/mL (non-virally suppressed) | 294 | 300 | 52 | 646
  Missing | 0 | 0 | 11 | 11

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Retained and Virally Suppressed Among Those Receiving the DTP Versus ICM Arms
Description: Retention and viral suppression at 18 months in those initially randomized to DTP vs. ICM. Participants are considered to be retained in care if they attended their 18-month final study visit and were engaged in care at 18-months. Viral suppression is defined as having less than 50 viral copies per milliliter.
Time Frame: 18 months after enrollment
Population: This outcome is presented as an intention to treat analysis based on baseline randomization (DTP vs. ICM). All 777 participants randomized at baseline are included here.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Decentralized Treatment Provision (DTP) at Baseline: DTP:
  * Standard of care, minus clinic referrals for ART treatment initiation and management.
  * Nurse initiated and managed ART within the community on mobile van at sites served by the mobile van which already provides SoC services
Arm/Group | Decentralized Treatment Provision (DTP) at Baseline | Individualized Case Management (ICM) at Baseline
Number analyzed (Participants) | 387 | 390
percentage of participants | 16.0 [12.4 to 19.7] | 14.1 [10.6 to 17.6]
Statistical Analysis 1: Comparison: Decentralized Treatment Provision (DTP) at Baseline vs Individualized Case Management (ICM) at Baseline; Test type: Superiority; p = 0.455, Two sample test of proportions — Threshold for significance: 0.05

2. Secondary Outcome: Retention and Viral Suppression of Non-Responders
Description: Retention and viral suppression at 18 months among month 6 non-responders randomized to continuation of either intervention vs. combined DTP+ICM
Time Frame: 18 months after enrollment
Population: This outcome was specified as a comparison of two subgroups rather than overall sample. This is why only two groups are included in this outcome and the number of participants is smaller than the total sample.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Rerandomized to Continue DTP or ICM if Non-responsive: DTP:
  * Standard of care, minus clinic referrals for ART treatment initiation and management.
  * Nurse initiated and managed ART within the community on mobile van at sites served by the mobile van which already provides SoC services
  OR
  ICM:
  * Standard of Care
  * Assignment of peer case manager
  * Face-to-face meeting to tailor ICM approach to FSW preference
  * Self-efficacy building in face-to-face sessions and bi-weekly text messages
  * Relational support through monthly calls, face-to-face meetings every three months, and additional support through FSW initiated interaction
- Rerandomized to Receive DTP+ICM if Non-responsive: DTP:
  * Standard of care, minus clinic referrals for ART treatment initiation and management.
  * Nurse initiated and managed ART within the community on mobile van at sites served by the mobile van which already provides SoC services
  AND
  ICM:
  * Standard of Care
  * Assignment of peer case manager
  * Face-to-face meeting to tailor ICM approach to FSW preference
  * Self-efficacy building in face-to-face sessions and bi-weekly text messages
  * Relational support through monthly calls, face-to-face meetings every three months, and additional support through FSW initiated interaction
Arm/Group | Rerandomized to Continue DTP or ICM if Non-responsive | Rerandomized to Receive DTP+ICM if Non-responsive
Number analyzed (Participants) | 351 | 328
percentage of participants | 11.4 [8.1 to 14.7] | 11.3 [7.9 to 14.7]
Statistical Analysis 1: Comparison: Rerandomized to Continue DTP or ICM if Non-responsive vs Rerandomized to Receive DTP+ICM if Non-responsive; Test type: Superiority; p = 0.962, Two sample test of proportions — Statistical significance threshold: 0.05

3. Secondary Outcome: Risk Factors of Loss to Follow-up
Description: Risk stratification to identify FSW at highest risk for loss to follow-up.
Time Frame: Up to 18 months after enrollment
Population: Risk factors for loss to follow up were analyzed across the sample, not by randomization assignment. Groups here reflect this approach.
Measure: Count of Participants; unit: Participants
Groups:
- Lost to Follow-up: Participants who were absent from any visits for 6 months or more.
- Not Lost to Follow-up (Retained in Care): Participants who attended a visit within the past 6 months
Arm/Group | Lost to Follow-up | Not Lost to Follow-up (Retained in Care)
Number analyzed (Participants) | 578 | 199
Participants
  Steady partner, living together | 87 | 36
  5 to 9 new clients in the past month | 159 | 40
  Marijuana use in the past 30 days | 227 | 66
  Experienced physical violence in the pasts 6 months | 338 | 103
  Experienced sexual violence in the past 6 months | 250 | 73
  Viral load of 50-1000 copies/mL at baseline | 130 | 54
  Viral load greater than 1000 copies/mL at baseline | 448 | 145
Statistical Analysis 1: Comparison: Lost to Follow-up vs Not Lost to Follow-up (Retained in Care); Statistical test for risk of LTFU for steady partner, living together vs. single; Test type: Superiority; p < 0.05, Regression, Cox — Threshold for statistical significance: 0.05; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.61 to 0.99]
Statistical Analysis 2: Comparison: Lost to Follow-up vs Not Lost to Follow-up (Retained in Care); Statistical test for risk of LTFU for 5-9 new clients in the past month vs. 0 clients in the past month; Test type: Superiority; p < 0.05, Regression, Cox — Threshold for statistical significance: 0.05; Hazard Ratio (HR) = 1.60, 95% CI 2-sided [1.02 to 2.51]
Statistical Analysis 3: Comparison: Lost to Follow-up vs Not Lost to Follow-up (Retained in Care); Statistical test for risk of LTFU for use of marijuana in the past 30 days vs. no marijuana use in the past 30 days; Test type: Superiority; p < 0.05, Regression, Cox — Threshold for statistical significance: 0.05; Hazard Ratio (HR) = 1.31, 95% CI 2-sided [1.09 to 1.57]
Statistical Analysis 4: Comparison: Lost to Follow-up vs Not Lost to Follow-up (Retained in Care); Statistical test for risk of LTFU among those experiencing physical violence in the past 6 months vs. no experience of physical violence in the past 6 months; Test type: Superiority; p < 0.05, Regression, Cox — Threshold for statistical significance: 0.05; Hazard Ratio (HR) = 1.24, 95% CI 2-sided [1.01 to 1.52]
Statistical Analysis 5: Comparison: Lost to Follow-up vs Not Lost to Follow-up (Retained in Care); Statistical test for risk of LTFU among those who have experienced sexual violence in the past 6 months vs. those who have not; Test type: Superiority; p < 0.05, Regression, Cox — Threshold for statistical significance: 0.05; Hazard Ratio (HR) = 1.62, 95% CI 2-sided [1.31 to 2.00]
Statistical Analysis 6: Comparison: Lost to Follow-up vs Not Lost to Follow-up (Retained in Care); Statistical test for risk of LTFU among those with viral loads from 50-1000 copies/mL at baseline vs. <50 copies/mL; Test type: Superiority; p < 0.05, Regression, Cox — Threshold for statistical significance: 0.05; Hazard Ratio (HR) = 2.33, 95% CI 2-sided [1.65 to 3.29]
Statistical Analysis 7: Comparison: Lost to Follow-up vs Not Lost to Follow-up (Retained in Care); Statistical test for risk of LTFU among those with viral load greater than 1000 copies/mL vs. those with viral load less than 50 copies/mL; Test type: Superiority; p < 0.05, Regression, Cox — Threshold for significance: 0.05; Hazard Ratio (HR) = 2.47, 95% CI 2-sided [1.82 to 3.36]

4. Secondary Outcome: Durability of Retention and Viral Suppression of Responders
Description: Durability of retention and viral suppression among 6 month responders continuing on DTP or ICM vs. those randomized to revert to standard of care (SoC)
Time Frame: Up to 18 months after enrollment
Population: This is a subgroup analysis of two of the month 6 re-randomization arms rather than the entire sample. Groups listed here and sample sizes reflect this approach.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- DTP or ICM, Continue DTP or ICM if Responsive: DTP:
  * Standard of care, minus clinic referrals for ART treatment initiation and management.
  * Nurse initiated and managed ART within the community on mobile van at sites served by the mobile van which already provides SoC services
  ICM:
  * Standard of Care
  * Assignment of peer case manager
  * Face-to-face meeting to tailor ICM approach to FSW preference
  * Self-efficacy building in face-to-face sessions and bi-weekly text messages
  * Relational support through monthly calls, face-to-face meetings every three months, and additional support through FSW initiated interaction
  Continues with intervention assigned at baseline (either DTP or ICM) if virally suppressed at 6 months.
- DTP or ICM, Standard of Care (SoC) if Responsive: DTP:
  * Standard of care, minus clinic referrals for ART treatment initiation and management.
  * Nurse initiated and managed ART within the community on mobile van at sites served by the mobile van which already provides SoC services
  ICM:
  * Standard of Care
  * Assignment of peer case manager
  * Face-to-face meeting to tailor ICM approach to FSW preference
  * Self-efficacy building in face-to-face sessions and bi-weekly text messages
  * Relational support through monthly calls, face-to-face meetings every three months, and additional support through FSW initiated interaction
  SoC:
  * HIV counseling and testing (HTC)
  * STI screening and treatment
  * TB screening and referral
  * Health education through peer educators and peer supported follow-up related to linkages to care
  * Referrals to DOH primary healthcare clinics or THC drop-in center for ART treatment initiation and management
  Returns to SoC if virally suppressed at 6 months.
Arm/Group | DTP or ICM, Continue DTP or ICM if Responsive | DTP or ICM, Standard of Care (SoC) if Responsive
Number analyzed (Participants) | 22 | 18
percentage of participants | 43.1 [29.5 to 56.7] | 40.0 [25.7 to 54.3]
Statistical Analysis 1: Comparison: DTP or ICM, Continue DTP or ICM if Responsive vs DTP or ICM, Standard of Care (SoC) if Responsive; Test type: Superiority; p = 0.756, Two sample test of proportions — Threshold of significance: 0.05

5. Secondary Outcome: Adherence Assessment
Description: Self-reported adherence to assess adherence across arms
Time Frame: 18 months
Population: This outcome was analyzed by baseline randomization status rather than month 6 re-randomization status. Groups included here reflect this. Numbers analyzed are smaller due to the fact that there was loss to follow up and not all participants answered questions on self-reported adherence.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Decentralized Treatment Provision (DTP) at Baseline | Individualized Case Management (ICM) at Baseline
Number analyzed (Participants) | 200 | 223
percentage of participants | 46.5 [39.6 to 53.4] | 51.6 [45.0 to 58.2]
Statistical Analysis 1: Comparison: Decentralized Treatment Provision (DTP) at Baseline vs Individualized Case Management (ICM) at Baseline; Test type: Superiority; p = 0.295, Two sample test of proportions — Threshold of statistical significance: 0.05

6. Secondary Outcome: Viral Suppression of Retained
Description: Among those retained, comparison of viral suppression across arms
Time Frame: Up to 18 months after enrollment
Population: This outcome was analyzed by baseline randomization status (DTP vs. ICM). Number of participants included reflects the total number retained in care across the two arms, which is less than the original sample size due to loss to follow up.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Decentralized Treatment Provision (DTP) at Baseline | Individualized Case Management (ICM) at Baseline
Number analyzed (Participants) | 214 | 231
percentage of participants | 29.0 [22.9 to 35.1] | 23.0 [17.6 to 28.4]
Statistical Analysis 1: Comparison: Decentralized Treatment Provision (DTP) at Baseline vs Individualized Case Management (ICM) at Baseline; Test type: Superiority; p = 0.149, Two sample test of proportions — Threshold for statistical significance: 0.05

7. Secondary Outcome: Loss-to-Follow-Up
Description: Loss-to-follow-up across arms (DTP vs. ICM). This outcome is presented as an intention to treat analysis based on baseline randomization (DTP vs. ICM). All 777 participants randomized at baseline are included here. Loss to follow-up is defined as having missed the 18-month final study visit.
Time Frame: 18 months after study enrollment
Population: This outcome was analyzed by baseline randomization assignment (DTP vs. ICM). Groups included here reflect this.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Decentralized Treatment Provision (DTP) at Baseline | Individualized Case Management (ICM) at Baseline
Number analyzed (Participants) | 387 | 390
percentage of participants | 45.0 [40.0 to 49.9] | 41.3 [36.4 to 46.2]
Statistical Analysis 1: Comparison: Decentralized Treatment Provision (DTP) at Baseline vs Individualized Case Management (ICM) at Baseline; Test type: Superiority; p = 0.301, Two sample test of proportions — Threshold of significance: 0.05

8. Secondary Outcome: Intervention Acceptability
Description: Participant reported intervention acceptability
Time Frame: Acceptability of each intervention at 6 month timepoint
Population: This outcome was analyzed by baseline randomization status (DTP vs. ICM) which is reflected in the two groups included here. The number for analysis is smaller than the overall sample due to not all participants responding to acceptability questions either due to refusal or loss to follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | Decentralized Treatment Provision (DTP) at Baseline | Individualized Case Management (ICM) at Baseline
Number analyzed (Participants) | 176 | 189
Participants | 163 | 156

9. Secondary Outcome: 2nd/3rd Line ART
Description: Number of participants who were tested and identified as resistant to first line therapy and were referred to a Department of Health facility for second line therapy across arms
Time Frame: Up to 18 months after enrollment
Population: This outcome was analyzed by baseline randomization as reflected in the two groups included. The number analyzed reflects the number of individuals who were tested for drug resistance which was a subset of the sample in line with protocol guidelines.
Measure: Count of Participants; unit: Participants
Arm/Group | Decentralized Treatment Provision (DTP) at Baseline | Individualized Case Management (ICM) at Baseline
Number analyzed (Participants) | 37 | 34
Participants | 36 | 32

10. Secondary Outcome: ART Resistance
Description: Report and compare resistance across arms
Time Frame: Up to 18 months after enrollment
Population: This outcome was analyzed by baseline randomization assignment as shown in the two groups included here. The number of participants analyzed represents those tested for drug resistance in line with protocol guidelines.
Measure: Count of Participants; unit: Participants
Arm/Group | Decentralized Treatment Provision (DTP) at Baseline | Individualized Case Management (ICM) at Baseline
Number analyzed (Participants) | 42 | 35
Participants | 37 | 34
Statistical Analysis 1: Comparison: Decentralized Treatment Provision (DTP) at Baseline vs Individualized Case Management (ICM) at Baseline; Test type: Superiority; p = 0.212, Chi-squared — Threshold of statistical significance: 0.05

11. Secondary Outcome: Participants' Costs South in African Rand (ZAR)
Description: Participants' cost data were collected by opportunity cost questionnaire for the intervention arms in the trial and are summarized descriptively to support potential future modeling. Participants' costs are defined as costs associated with attending each visit for HIV care (transportation, food, child-care and other; and money that would have been earned from clients (opportunity cost). Follow-up costs were for attending each DTP/ICM and HIV care clinic visit.
Time Frame: Baseline, Follow-up up to 5 months
Population: Participants with cost questionnaire data collected were included in analyses.
Measure: Mean (Inter-Quartile Range); unit: ZAR
Groups:
- Decentralized Treatment Provision (DTP): DTP:
  Standard of care, minus clinic referrals for ART treatment initiation and management.
  Nurse initiated and managed ART within the community on mobile van at sites served by the mobile van which already provides SoC services
- Individualized Case Management (ICM): ICM:
  Standard of Care Assignment of peer case manager Face-to-face meeting to tailor ICM approach to FSW preference Self-efficacy building in face-to-face sessions and bi-weekly text messages Relational support through monthly calls, face-to-face meetings every three months, and additional support through FSW initiated interaction
Arm/Group | Decentralized Treatment Provision (DTP) | Individualized Case Management (ICM)
Number analyzed (Participants) | 183 | 176
ZAR
  Baseline | 186.8 [21.5 to 250] | 164.9 [12 to 233]
  Follow-up up to 5 months: number analyzed (Participants) | 34 | 22
  Follow-up up to 5 months | 127.7 [0 to 137.5] | 256.1 [34.3 to 361.8]

12. Other Pre Specified Outcome: Decentralized Treatment Provision (DTP) Pick-Ups
Description: Number and percentage of DTP pick-ups attended among participants randomized to received DTP.
Time Frame: Up to 18 months after enrollment
Population: Only a subset of participants received the DTP intervention either from baseline or at 6 months (550 total). The number of units represents the total expected number of DTP pickups per protocol.
Measure: Count of Units; unit: Total DTP pickups
Units Other Than Participants: Total DTP pickups
Groups:
- Decentralized Treatment Provision (DTP) at Baseline and/or 6 Months: DTP:
  * Standard of care, minus clinic referrals for ART treatment initiation and management.
  * Nurse initiated and managed ART within the community on mobile van at sites served by the mobile van which already provides SoC services
Arm/Group | Decentralized Treatment Provision (DTP) at Baseline and/or 6 Months
Number analyzed (Participants) | 550
Number analyzed (Total DTP pickups) | 8634
Total DTP pickups | 3332

13. Other Pre Specified Outcome: ICM Phone-Based Contacts
Description: Number of ICM phone-based contacts
Time Frame: Up to 18 months after enrollment
Population: Only a subset of participants received the ICM intervention, either from baseline or at 6 months (552 total). The units analyzed represent the total number of expected phone calls per protocol.
Measure: Count of Units; unit: Planned phone-based contacts
Units Other Than Participants: Planned phone-based contacts
Groups:
- Individualized Case Management (ICM) at Baseline and/or 6 Months: ICM:
  * Standard of Care
  * Assignment of peer case manager
  * Face-to-face meeting to tailor ICM approach to FSW preference
  * Self-efficacy building in face-to-face sessions and bi-weekly text messages
  * Relational support through monthly calls, face-to-face meetings every three months, and additional support through FSW initiated interaction
Arm/Group | Individualized Case Management (ICM) at Baseline and/or 6 Months
Number analyzed (Participants) | 552
Number analyzed (Planned phone-based contacts) | 8640
Planned phone-based contacts | 593

14. Other Pre Specified Outcome: ICM In-Person Meetings
Description: Percentage of face-to-face case manager sessions attended
Time Frame: Up to 18 months after enrollment
Population: Only a subset of participants received the ICM intervention, either from baseline or at month 6 (552 total). The units analyzed represent the number of expected in person sessions per protocol.
Measure: Count of Units; unit: Number of planned in-person ICM sessions
Units Other Than Participants: Number of planned in-person ICM sessions
Arm/Group | Individualized Case Management (ICM) at Baseline and/or 6 Months
Number analyzed (Participants) | 552
Number analyzed (Number of planned in-person ICM sessions) | 1273
Number of planned in-person ICM sessions | 392

ADVERSE EVENTS:
Time Frame: Up to 18 months
Description: AEs were systematically investigated during lost to follow up tracing. Recent experiences of physical and sexual violence, hospitalizations were captured at study visits. All AEs were reported to the data safety & monitoring board 6-monthly and institutional review board annually. None of the AEs, SAEs, or deaths reported were related to study involvement.
  AEs are reported by baseline randomization status in line with how they were systematically followed up on and documented by the two arms.
Groups:
- Decentralize Treatment Provision (DTP) at Baseline: DTP:
  * Standard of care, minus clinic referrals for ART treatment initiation and management.
  * Nurse initiated and managed ART within the community on mobile van at sites served by the mobile van which already provides SoC services
- Standard of Care (SoC) at Baseline: SoC:
  * HIV counseling and testing (HTC)
  * STI screening and treatment
  * TB screening and referral
  * Health education through peer educators and peer supported follow-up related to linkages to care
  * Referrals to DOH primary healthcare clinics or THC drop-in center for ART treatment initiation and management
  Returns to SoC if virally suppressed at 6 months.
  ICM: Peer-led ICM through quarterly face-to-face meetings, monthly phone calls and biweekly text messages.
- Enrolled But Not Randomized: A subset of participants were enrolled in the study but not randomized for the following reasons:
  * Missing viral loads (unknown viral suppression status)
  * Unable to randomize due to losing contact after enrollment
  * Mistakenly put in standard of care group (protocol violation)
  * Withdrew from study
Arm/Group | Decentralize Treatment Provision (DTP) at Baseline | Individualized Case Management (ICM) at Baseline | Standard of Care (SoC) at Baseline | Enrolled But Not Randomized
All-Cause Mortality (participants affected / at risk) | 4/387 | 12/390 | 1/523 | 0/91
Serious Adverse Events (participants affected / at risk) | 8/387 | 16/390 | 1/523 | 0/91
Other Adverse Events (participants affected / at risk) | 0/387 | 0/390 | 0/523 | 0/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Decentralize Treatment Provision (DTP) at Baseline (N=387) | Individualized Case Management (ICM) at Baseline (N=390) | Standard of Care (SoC) at Baseline (N=523) | Enrolled But Not Randomized (N=91)
Imprisoned while enrolled in study (Social circumstances) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Physical violence (Social circumstances) | 1 (1) | 3 (3) | 0 (0) | 0 (0) — Experienced physical violence while enrolled in study (unrelated to study participation)
Hospitalization (Social circumstances) | 3 (3) | 3 (3) | 1 (1) | 0 (0) — Hospitalization during enrollment unrelated to study participation
Motor vehicle accident (Social circumstances) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Stroke (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Not related to study participation
Gallstones and swollen feet (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Not related to study participation
Sexual violence (Social circumstances) | 1 (1) | 4 (4) | 0 (0) | 0 (0) — Not related to study participation

LIMITATIONS AND CAVEATS:
A limitation to this study has been determining engagement in care and viral load status for those who were lost to follow up (LTFU) in the trial in order to inform the primary outcome. Given the high rates of LTFU, participants may have been seeking care elsewhere and achieved viral suppression during the follow up period without our knowledge. This has implications for our primary outcome which uses an intention to treat (ITT) analysis of engagement in care and viral suppression.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-04-09): https://cdn.clinicaltrials.gov/large-docs/72/NCT03500172/Prot_SAP_002.pdf
  • Informed Consent Form (2018-04-04): https://cdn.clinicaltrials.gov/large-docs/72/NCT03500172/ICF_004.pdf